CLINICAL TRIAL: NCT05233839
Title: The Effect of Telerehabilitation and Conventional Rehabilitation on Clinical Outcomes and Exercise Compliance in Patients With Degenerative Meniscal Injury
Brief Title: Efficacy of Telerehabilitation in Patients With Degenerative Meniscal Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mugla
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Meniscus; Degeneration
Keywords: Degenerative meniscus injury; Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) (Experimental): The TR group will be followed up through the application within the 8-week home exercise program.
  Interventions: Other: Telerehabilitation
- Paper Based Rehabilitation (PBR) (Active Comparator): The PBR group will be followed up through the paper instruction within the 8-week home exercise program.
  Interventions: Other: Paper Based Rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Application based video home exercise for the degenerative meniscus injury
  Arms: Telerehabilitation (TR)
Other: Paper Based Rehabilitation — Paper instruction based home exercise for the degenerative meniscus injury
  Arms: Paper Based Rehabilitation (PBR)

SUMMARY:
The aim of the study is to compare the home exercise program performed with video-based telerehabilitation in patients with degenerative meniscal injury, and the home exercise program performed with one-on-one training in the hospital with conventional methods.

DETAILED DESCRIPTION:
Conventional rehabilitation (CR) practices will be applied to the first study group. Telerehabilitation (TR) application will be applied to the second study group. It is aimed to evaluate the patients in terms of pain, functionality, quality of life and exercise compliance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 - 65 years
* Having been diagnosed with degenerative meniscus injury by an orthopedist by MRI examination
* Having signed the consent form

Exclusion Criteria:

* Situations that will prevent assessments or communication with the individual
* Having an operation due to degenerative meniscus injury problem
* Orthopedic and neurological problems that would prevent evaluation and/or treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numerical scale (0: no pain, 10: unbearable pain).
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 8 weeks
  WOMAC consists of 3 main headings: pain intensity, stiffness, and physical function. The total score ranges from 0 (no disability) to 96 (complete disability).
SF-12 | Change from Baseline SF-12 at 8 weeks
  SF 12 is a self-evaluation scale. It consists of seven items. Its score ranged from 0 to 100, with higher scores indicating better physical and mental health functioning.
Muscle Strength Test with Lafayette Hand Held Dynamometer | Change from Baseline Dynamometer Value at 8 weeks
  It is an objective muscle strength measurement tool. Measurements are made 3 times. A rest of 120 seconds is given between measurements. The highest measured value is noted.
Proprioception Measurement with Baseline Bubble Inclinometer | Change from Baseline Inclinometer Value at 8 weeks
  The "absolute angle difference", which is the difference between the targeted angle and the angle realized by the patient in each repetition, is recorded. The arithmetic mean of the absolute angle difference of 3 repetitions is the result data.

SECONDARY OUTCOMES:
EARS | Change from Baseline EARS at 8 weeks
  In order to observe the individual's adaptation to exercise, the motivation levels of the patients regarding the exercise program are evaluated with the exercise diary prepared by the researchers of the study. It is scored between 0 to 24. Higher scores indicate greater adherence.
TSUQ | Change from Baseline TSUQ at 8 weeks
  It consists of 21 items. With this survey, the satisfaction levels and usability of individuals using the telemedicine service are evaluated. The total score is scored between 17 and 85. Higher scores indicate higher satisfaction and usability.

CONTACTS AND LOCATIONS:
Overall Officials: İsmet Tümtürk, BSc, Principal Investigator — Ege University; Cem Yalın Kılınç, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No